CLINICAL TRIAL: NCT01936311
Title: Study of Screening for Patients Self-selected Health Goal and Treatment Modality Prior to Primary Care Visit and the Effect on Short-term Behavior Change
Brief Title: Study of Screening Self-management Goals on Short Term Behavior Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: Advancing Care Together (Unknown); Colorado Health Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHF-3848; 13-1523 (Other: COMIRB)
Record Dates: First submitted 2013-09-03; First posted 2013-09-06 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Patient Health Behaviors
Keywords: Health Behavior; Behavior change; self-management goal; health goal
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): This group will receive usual care.
- Self-Management Goal Elicitation (Experimental): This group will receive usual care alongside a form that helps elicit self-management goals as well as preferred treatment modalities.
  Interventions: Behavioral: Self-management goal elicitation

INTERVENTIONS:
Behavioral: Self-management goal elicitation — The intervention will be a form, given prior to a primary care visit, that allows patients to express a self-management goal (health goal) they would like to work on, and a preferred treatment modality.
  Arms: Self-Management Goal Elicitation

SUMMARY:
The purpose of this study is to test whether having patients identify a self-management goal (health goal), prior to a visit with their primary care provider, leads to health behavior improvement over six weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years of age)
* Attending primary care visit at Lowry Family Health Center or Level One Physicians
* English- or Spanish-Speaking

Exclusion Criteria:

* Exhibit signs of cognitive impairment or significant hearing impairment
* Provider recommendation against enrolling in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2013-06; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Self-rated health | 6 weeks
  Single item measure of self rated health:
  "How would you rate your overall health during the past week? (1=Very Poor, 7=Excellent)?"
  We will compare scores between groups as well as change over 6-weeks between groups.

SECONDARY OUTCOMES:
Health behavior improvement | 6 Weeks
  Our secondary outcome measure will include a measure of behavior specific improvements. We will evaluate both component improvements for their specified behavior, as well as the composite score of negative health behaviors assessed from a series of questions.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Level One Physicians, Denver, Colorado
  - Lowry Family Health Center, Denver, Colorado